CLINICAL TRIAL: NCT05187598
Title: Evaluation of the Effectiveness of Online Communication Training Focused on Maintaining Perinatal Patient Safety for Nursing Students
Brief Title: The Effect of Communication Training on the Communication Skills of the Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Cigdem Yucel Ozcırpan (Unknown); Sergul Duygulu (Unknown)
Responsible Party: Principal Investigator, SEVDA YILDIRIM HAMURCU, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GO 19/74
Record Dates: First submitted 2021-12-20; First posted 2022-01-12 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Communication, Multidisciplinary
Keywords: nursing students; communication; patient safety; standard participant
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: parallel group randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor does not know who is in the control group and who is in the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effective communication training in perinatal patient safety (Experimental): Nursing department students will be given training on effective communication training in perinatal patient safety.
  Interventions: Other: Effective communication training in perinatal patient safety
- Control group (No Intervention): There is no intervention for this group

INTERVENTIONS:
Other: Effective communication training in perinatal patient safety — Students will be given theoretical training, group discussion will be made over sample videos, and students will participate in the standard participant practice and a post-analysis session will be held.
  Arms: Effective communication training in perinatal patient safety

SUMMARY:
Patient safety, which is an important concept in terms of providing effective and high-quality health care, is defined as "preventing health care errors and eliminating or reducing patient damage caused by health care errors". Worldwide, adverse events from unsafe care are estimated to be one of the 10 leading causes of death and disability. Ineffective communication between healthcare professionals, which is among the factors that cause errors related to patient safety, is reported as one of the factors that have the most impact on medical errors and unintentional patient harm. Studies show that ineffective communication between healthcare professionals may be responsible for up to 80% of all preventable adverse events rather than the patient's medical condition. Considering the number of lawsuits and cost increase due to errors that violate patient safety, it is stated that medical errors are higher especially in the field of perinatology. In studies conducted, errors in the communication process were identified as the main cause in 72% of all perinatal deaths. The perinatal period is a physiological process. However, undesirable events can develop suddenly and rapidly, and this situation threatens both pregnant/mother and fetus/newborn health. Therefore, it is necessary to maintain uninterrupted communication in this area. It is very important for students to acquire these communication skills effectively before they graduate. Therefore, this research; In order to determine the effect of professional communication training among health professionals to be given to nursing students on the professional communication skills of students, a parallel-group was planned as a randomized controlled trial. The study is planned to be conducted in Hacettepe University Nursing Faculty. Research data will be collected using the Student Introductory Information Form, Effective Communication Skills Among Healthcare Professionals Evaluation Form, Self-Assessment Form for Effective Communication among Healthcare Professionals, and Semi-Structured Focus Group Interview Form. Nursing students who meet the inclusion criteria will be included in the research. Students will be divided into 2 groups as the experimental and the control group. Students in the experimental group will be given training on effective communication among health professionals. No training will be given to the control group.

ELIGIBILITY:
Inclusion Criteria:

* To have taken the course of Obstetrics-Gynecology Nursing,
* To be able to understand, and speak Turkish at a good level,
* Being able to use a computer,
* Having personal internet access.
* To be a volunteer.

Exclusion Criteria:

* Not participating in any stage of the research,
* Having a disability (physical/visual/auditory) that may prevent computer and internet use,
* Wanting to leave the at any stage of the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Effective communication form among perinatal healthcare professionals | 1 week before the intervention to 1 week after the intervention.
  It is the evaluation of the professional communication of nursing students with a nurse and a physician working in the perinatal area through an effective communication form.
Self-assessments of effective communication skills form among perinatal healthcare professionals | 1 week before the intervention to 1 week after the intervention.
  It is the self-evaluation of nursing students for their professional communication with a nurse and a physician working in the perinatal area through an effective communication self-assessment form.

CONTACTS AND LOCATIONS:
Overall Officials: Sergul Duygulu, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD
Supporting Information: Study Protocol
Time Frame: December 2022
Access Criteria: Statistical analyzes of the study will be made by an expert. The data will be shared with the expert by providing statistical blinding. The results of the study will be published in an international journal.

REFERENCES:
- [Background] Janakiraman V, Ecker J. Quality in obstetric care: measuring what matters. Obstet Gynecol. 2010 Sep;116(3):728-732. doi: 10.1097/AOG.0b013e3181ea4d4f. PMID 20733459
- [Background] Deering S, Johnston LC, Colacchio K. Multidisciplinary teamwork and communication training. Semin Perinatol. 2011 Apr;35(2):89-96. doi: 10.1053/j.semperi.2011.01.009. PMID 21440817
- [Background] Hailu FB, Kassahun CW, Kerie MW. Perceived Nurse-Physician Communication in Patient Care and Associated Factors in Public Hospitals of Jimma Zone, South West Ethiopia: Cross Sectional Study. PLoS One. 2016 Sep 15;11(9):e0162264. doi: 10.1371/journal.pone.0162264. eCollection 2016. PMID 27632162
- [Background] Hogan H, Zipfel R, Neuburger J, Hutchings A, Darzi A, Black N. Avoidability of hospital deaths and association with hospital-wide mortality ratios: retrospective case record review and regression analysis. BMJ. 2015 Jul 14;351:h3239. doi: 10.1136/bmj.h3239. PMID 26174149
- [Background] James JT. A new, evidence-based estimate of patient harms associated with hospital care. J Patient Saf. 2013 Sep;9(3):122-8. doi: 10.1097/PTS.0b013e3182948a69. PMID 23860193
- [Background] Jha AK, Prasopa-Plaizier N, Larizgoitia I, Bates DW; Research Priority Setting Working Group of the WHO World Alliance for Patient Safety. Patient safety research: an overview of the global evidence. Qual Saf Health Care. 2010 Feb;19(1):42-7. doi: 10.1136/qshc.2008.029165. PMID 20172882
- [Background] Karkowsky CE, Chazotte C. Simulation: improving communication with patients. Semin Perinatol. 2013 Jun;37(3):157-60. doi: 10.1053/j.semperi.2013.02.006. PMID 23721771
- [Background] Leonard M, Graham S, Bonacum D. The human factor: the critical importance of effective teamwork and communication in providing safe care. Qual Saf Health Care. 2004 Oct;13 Suppl 1(Suppl 1):i85-90. doi: 10.1136/qhc.13.suppl_1.i85. PMID 15465961
- [Background] Lippke S, Derksen C, Keller FM, Kotting L, Schmiedhofer M, Welp A. Effectiveness of Communication Interventions in Obstetrics-A Systematic Review. Int J Environ Res Public Health. 2021 Mar 5;18(5):2616. doi: 10.3390/ijerph18052616. PMID 33807819
- [Background] Lyndon A. Communication and teamwork in patient care: how much can we learn from aviation? J Obstet Gynecol Neonatal Nurs. 2006 Jul-Aug;35(4):538-46. doi: 10.1111/j.1552-6909.2006.00074.x. PMID 16882000
- [Background] Makary MA, Daniel M. Medical error-the third leading cause of death in the US. BMJ. 2016 May 3;353:i2139. doi: 10.1136/bmj.i2139. No abstract available. PMID 27143499
- [Background] Martinez-Galiano JM, Martinez-Vazquez S, Rodriguez-Almagro J, Hernandez-Martinez A. The magnitude of the problem of obstetric violence and its associated factors: A cross-sectional study. Women Birth. 2021 Sep;34(5):e526-e536. doi: 10.1016/j.wombi.2020.10.002. Epub 2020 Oct 17. PMID 33082123
- [Background] Muller M, Jurgens J, Redaelli M, Klingberg K, Hautz WE, Stock S. Impact of the communication and patient hand-off tool SBAR on patient safety: a systematic review. BMJ Open. 2018 Aug 23;8(8):e022202. doi: 10.1136/bmjopen-2018-022202. PMID 30139905
- [Background] Pettker CM, Thung SF, Lipkind HS, Illuzzi JL, Buhimschi CS, Raab CA, Copel JA, Lockwood CJ, Funai EF. A comprehensive obstetric patient safety program reduces liability claims and payments. Am J Obstet Gynecol. 2014 Oct;211(4):319-25. doi: 10.1016/j.ajog.2014.04.038. Epub 2014 Jun 9. PMID 24925798
- [Background] Reising DL, Carr DE, Gindling S, Barnes R, Garletts D, Ozdogan Z. Team Communication Influence on Procedure Performance: Findings From Interprofessional Simulations with Nursing and Medical Students. Nurs Educ Perspect. 2017 Sep/Oct;38(5):275-276. doi: 10.1097/01.NEP.0000000000000168. PMID 28562460
- [Background] Vincent C, Amalberti R. Safety in healthcare is a moving target. BMJ Qual Saf. 2015 Sep;24(9):539-40. doi: 10.1136/bmjqs-2015-004403. Epub 2015 Jul 6. No abstract available. PMID 26150547
- [Background] Woloshynowych M, Rogers S, Taylor-Adams S, Vincent C. The investigation and analysis of critical incidents and adverse events in healthcare. Health Technol Assess. 2005 May;9(19):1-143, iii. doi: 10.3310/hta9190. PMID 15890139
- [Background] Zavertnik JE, Huff TA, Munro CL. Innovative approach to teaching communication skills to nursing students. J Nurs Educ. 2010 Feb;49(2):65-71. doi: 10.3928/01484834-20090918-06. Epub 2010 Feb 4. PMID 19810670